CLINICAL TRIAL: NCT00399633
Title: Neuropeptides in the Humane Intra- og Extracerebral Circulation - in Relation to Sumatriptan in Healthy Volunteers.
Brief Title: Neuropeptides in the Humane Intra- og Extracerebral Circulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Bispebjerg Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: Neuropeptide2007
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Healthy; Migraine
Keywords: VIP; PACAP; CGRP; Prostanoids
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

INTERVENTIONS:
Drug: sumatriptan

SUMMARY:
The study aim at examining whether Sumatriptan changes the plasma values of the neuropeptides vasoactive intestinal polypeptide (VIP), calcitonin gene-related peptide (CGRP) and pituitary adenylate cyclase activating peptide (PACAP) and the prostanoids 6-keto-PGF1α, and PGE2, PGD2 og PGF2α.

DETAILED DESCRIPTION:
The study is meant to give a better understanding of the basic mechanisms behind migraine, and a better understanding of the effects of sumatriptan on the trigemino vascular system.

The endpoints are changes in the plasma values of the neuropeptides vasoactive intestinal polypeptide (VIP), calcitonin gene-related peptide (CGRP) and pituitary adenylate cyclase activating peptide (PACAP) and the prostanoids 6-keto-PGF1α, and PGE2, PGD2 og PGF2α.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* 18-50 years,
* 50-100 kg.
* Fertile women must use birth control.

Exclusion Criteria:

* All primary types of headache
* Daily intake of medicine except birth control
* Pregnancy
* Hypertension
* Hypotension
* other chronic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Blood concentration of vasoactive intestinal polypeptide (VIP),
calcitonin gene-related protein (CGRP), pituitary adenylate cyclase
activating peptide (PACAP,) and the prostanoids
6-keto-PGF1α, PGE2, PGD2 and PGF2α, sampled from different
venous catheters.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup, Copenhagen, Copenhagen, Denmark